CLINICAL TRIAL: NCT07387835
Title: The Effect of Rhythm-Based Stabilization Training on Scapular Control, Upper Extremity Performance, and Range of Motion in Video Gamers.
Brief Title: Rhythm-Based Stabilization Training in Video Gamers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Ali Wakid, Principal Investigator, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-392
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Scapular Dyskinesis; Shoulder Pain; Postural Impairment
Keywords: Video Gamers; Rhythmic Stabilization; Scapular Control; Neuromuscular Training; Upper Extremity Performance
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): This group will receive a 4-week rhythm-based scapular stabilization program consisting of 6 specific exercises performed twice weekly. The protocol combines exercises on stable and unstable surfaces to enhance neuromuscular control and scapular stability.
  Interventions: Other: Rhythm-Based Scapular Stabilization Program
- Control Group (Other): Following the assessment session, posture training and general information will be provided. Participants in this group will not participate in the stabilization exercise program. They will be instructed to maintain their regular daily activities and gaming routines without any specific therapeutic intervention during the 4-week study period.
  Interventions: Other: Posture education

INTERVENTIONS:
Other: Rhythm-Based Scapular Stabilization Program — "A 4-week exercise program consisting of 6 specific scapular stabilization exercises based on the rhythmic stabilization technique. The program includes 2 sets of 10 repetitions for each exercise, performed twice weekly. It utilizes both stable surfaces (wall/table) and unstable surfaces (Swiss balls) to challenge neuromuscular control and improve scapular stability in video gamers."
  Arms: Experimental Group
Other: Posture education — Posture education and general information
  Arms: Control Group

SUMMARY:
This study aims to evaluate the effectiveness of a 4-week rhythm-based stabilization exercise protocol for professional video gamers diagnosed with scapular dyskinesis. Participants will undergo a structured exercise program consisting of 6 specific scapular stabilization exercises. These exercises will be performed on both stable surfaces (such as a treatment table or wall) and unstable surfaces (such as Swiss balls) to challenge neuromuscular control. The primary goal is to determine how this combined approach affects scapular control, upper extremity functional performance, and joint range of motion. Data will be collected through clinical assessments before and after the 4-week intervention to measure improvements in scapular stability and overall upper limb function.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participants between 18 and 35 years of age
* Playing video games for at least 3 hours per week for at least 3 months.
* Healthy individuals with no chronic or acute shoulder/upper extremity problems.
* Not participated in any other upper extremity treatment program in the last 6 months.
* Willingness to participate and sign the informed consent form

Exclusion Criteria:

* History of trauma, surgery, or fracture in the shoulder, neck, or hand in the last 6 months.
* Diagnosis of any neurological disease (e.g., MS, Stroke).
* Structural causes of upper extremity pain, such as disc herniation or radiculopathy.
* Vestibular or balance disorders affecting upper extremity movement
* Inability to perform required exercises due to severe pain or physical limitations

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
Upper Quarter Closed Kinetic Chain Stability Test (UQCKCST) | 4 weeks
  This is a low-cost test that evaluates the functional performance and stability of the upper extremity in a closed kinetic chain. For the test, the participant assumes a push-up position with their hands placed 90 cm apart; men use the full position, while women use a modified (knees on the ground) position. The test is based on the principle of touching one hand to the other as quickly as possible within 15 seconds and returning to the starting position, and the total number of touches is recorded as a score. The participant performs three trials separated by 45-second rest periods.
Reaction Time | 4 weeks
  Reaction Time is used to assess upper extremity reaction time and motor speed in athletes and young adults. In this study, a visual-cognitive reaction technology device (Blazepod) that has been shown to have high reliability will be used. Participants will be asked to turn off the light pods, which are randomly placed on the ground, by touching them with their dominant hand as quickly as possible when they are turned on. During the application, each participant will perform 5 trials separated by a 5-second rest period. Measurements will be recorded in milliseconds (ms), excluding the fastest and slowest values, and the average reaction time will be recorded.
Lateral Scapular Shift Test | 4 weeks
  This is a static test used to assess scapular asymmetry and medial-lateral inferior angle displacement. The measurement is taken by measuring the distance between the inferior angle of the scapula and the corresponding thoracic spine process with a tape measure while the participant is standing upright. The test is performed in three different arm positions:
  * Arm in neutral position, free at the sides.
  * Arm in 45° abduction, hands on hips.
  * Arm in 90° abduction, hands above the head (or thumbs pointing upwards). A difference of more than 1.5 cm between the right and left sides is considered clinically significant scapular asymmetry.
Scapular Muscle Endurance Test | 4 weeks
  This test is performed in a standing position to measure the endurance of the scapular stabilizing muscles. The participant stabilizes their scapula in a neutral position with their shoulder and elbow flexed at 90°, and maintains a 1 kg load determined by a dynamometer. The test continues until the participant can no longer maintain the position or the load. The measurement is repeated twice, and the longest time achieved is recorded in seconds.
Upper Quarter Y-Balance Test (YBT-UQ) | 4 weeks
  It is a tool developed to assess upper extremity performance and overall upper trunk stability at the limits. The test aims to identify movement limitations and asymmetries in pre-sports and rehabilitation screening. The participant assumes a push-up position with one hand placed on a support platform and attempts to reach the furthest possible distance with the other hand in 3 different directions: medial (inner), inferolateral (downward-outward), and superolateral (upward-outward). Attempts must be completed without losing balance or moving the standing hand.
Wrist Range of Motion (ROM) | 4 weeks
  Joint range of motion is a crucial component of upper extremity functional performance. This study will evaluate wrist flexion/extension and radial/ulnar deviation movements, as well as finger flexion/extension movements. Measurements will be taken using the HandROM Measurement System, which has been shown to be a reliable alternative to traditional goniometers. The system will allow for objective analysis of upper extremity functions, scapular control, and hand performance.
Medicine Ball Throw Test | 4 weeks
  This test will be used to evaluate upper extremity explosive power. Participants position themselves upright in a chair without armrests, with their ankles, knees, and hips at a 90-degree angle. They are then asked to grasp a 3 kg medicine ball with both hands and throw it forward overhead without leaning forward or flexing their elbows. The point where the ball first touches the ground is measured from the starting point and recorded in centimeters.

SECONDARY OUTCOMES:
Visual Analog Scale | 4 weeks
  The Visual Analog Scale will be used to assess the subjective intensity of pain experienced by the participant. This scale is a validated self-assessment tool for acute and chronic pain, rated from 0 ("no pain") to 10 ("unbearable pain"). Participants will be asked to rate the severity of their pain, particularly in the shoulder and upper extremity region, within this range.
The Shoulder Pain and Disability Index | 4 weeks
  The Shoulder Pain and Disability Index is a 13-item self-report questionnaire developed to assess the severity of shoulder pain and associated functional limitations in patients.The questionnaire includes a Pain subsection consisting of 5 items and a Disability subsection consisting of 8 items. Participants are asked to rate each item on a numerical rating scale (NRS) from 0 to 10. The validity and reliability of the questionnaire in Turkish have been proven. The final result is calculated as a percentage out of 100; a higher score indicates greater pain and disability.

IPD SHARING:
Plan to Share IPD: No